CLINICAL TRIAL: NCT02981537
Title: Two-staged Approach in Positioning Endobronchial Blockers Without Fiberoptic Guidance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jae-Hyon Bahk, MD, PhD, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: JHBahk_blocker
Record Dates: First submitted 2016-12-01; First posted 2016-12-05 (Estimated); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: One-lung Ventilation

ARMS (2):
- two-staged (Experimental): positioning endobronchial blockers to appropriate bronchus with two-staged methods
  Interventions: Device: two-staged endobronchial blocker insertion; Device: single-staged endobronchial blocker insertion
- single-staged (Active Comparator): positioning endobronchial blockers with traditional single-staged methods
  Interventions: Device: two-staged endobronchial blocker insertion; Device: single-staged endobronchial blocker insertion

INTERVENTIONS:
Device: two-staged endobronchial blocker insertion — positioning endobronchial blockers in two-staged method
Device: single-staged endobronchial blocker insertion — positioning endobronchial blockers in traditional single-staged method

SUMMARY:
The purpose of this study is to find a novel method for placing endobronchial blockers without fiberoptic guidance to provide one-lung isolation during anesthesia for thoracic surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for lung resection

Exclusion Criteria:

* refuse to enroll
* patients with lesions involving mainstem bronchi
* patients with anomalies in tracheobronchial tree

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2016-10; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
location of endobronchial blocker | immediately after the insertion of blocker by fiberoptic bronchoscope

CONTACTS AND LOCATIONS:
Overall Officials: JH Bahk, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Min S, Yoon S, Han J, Seo JH, Bahk JH. A novel technique of blindly positioning bronchial blockers for one-lung ventilation: a prospective, randomized, crossover study. J Cardiothorac Surg. 2025 Jan 9;20(1):50. doi: 10.1186/s13019-024-03276-8. PMID 39780264